CLINICAL TRIAL: NCT04554316
Title: Aesthetic Effect of Steri-Strip Orientation on Healing and Scar Appearance in Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, Candace Ward, Principal Investigator, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB-2019-118
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Scar; Breast Neoplasms; Breast Diseases; Surgical Wound
Keywords: wound healing; cosmesis; postoperative dressing
MeSH Terms: conditions — Cicatrix; Breast Neoplasms; Breast Diseases; Surgical Wound

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Parallel placement (Active Comparator): Steri-strips will be placed in-line (parallel) with the surgical incision.
  Interventions: Device: Steri-strip
- Perpendicular placement (Active Comparator): Steri-strips will be placed perpendicular to the surgical incision.
  Interventions: Device: Steri-strip

INTERVENTIONS:
Device: Steri-strip — Steri-Strips (3M Health Care, St. Paul, Minn) are a commonly used means of covering surgical incisions following many operations. Use of adhesive surgical tape over incisions maintains epidermal approximation in primary skin closure while limiting exposure to the environment, theoretically improving cosmesis and limiting risk of infection.

SUMMARY:
All patients undergoing breast biopsy, lumpectomy, needle-localization-guided breast biopsy, and mastectomy at Einstein Medical Center Philadelphia, Einstein Medical Center Montgomery, Center One, or Einstein Elkins Park will be offered participation into the study. Patients who have documented allergies to adhesive or tape, patients taking chronic steroids, and patients with documented connective tissue, skin, or healing disorders will be excluded from the study. Risks and benefits of the study as well as risks and benefits of the procedure will be discussed with the patient by one of the investigators. If the patient elects to participate in the study, they will be assigned to incisional dressing at the time of operation with either in-line or perpendicular placement of Steri-Strips based on the patient's computer-generated randomization assignment. The patient's chart will be reviewed to determine the patient's age and comorbid conditions including obesity (pre-operative BMI), diabetes mellitus, use of anti-platelet or anticoagulant medication, or smoking. This information will be utilized to ensure that our study groups are similar in baseline demographics and pre-existing conditions. Additionally, the primary medical reason for needing breast surgery will be reviewed as well as treatment with pre-operative or post-operative chemotherapy or radiation therapy to the breast. Steri-Strips will not be removed and will be allowed to fall off naturally. At regularly scheduled 30-day and 90-day follow-up appointments, pictures will be taken of the incisional area. These photographs will be reviewed by a blinded, independent surgeon who will grade each incision according to the modified Hollander Cosmesis Scale. Statistical analysis with t-testing of the means and chi-squared testing of dichotomous variables will be performed to determine significance of the findings.

ELIGIBILITY:
Inclusion Criteria:

- All adult patients undergoing breast biopsy, lumpectomy, needle-localization-guided breast biopsy, and mastectomy at Einstein Medical Center Philadelphia, Einstein Medical Center Montgomery, Center One, or Einstein Medical Center Elkins Park will be offered participation into the study.

Exclusion Criteria:

* Patients who have documented allergies to adhesive or tape, patients taking chronic steroids, and patients with documented connective tissue, skin, or healing disorders
* members of vulnerable populations such as adults who are unable to consent, individuals who are not yet adults, pregnant women, or prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Cosmesis score 30 days | 30 days
  Hollander cosmesis scale (0-6, 6 being best cosmetic grade) grade of scar appearance at 30 days
Cosmesis score 90 days | 90 days
  Hollander cosmesis scale (0-6, 6 being best cosmetic grade) grade of scar appearance at 90 days

SECONDARY OUTCOMES:
Surgical site infection | 90 days
  Presence or absence of surgical site infection
Wound dehiscence | 90 days
  Presence or absence of wound dehiscence

CONTACTS AND LOCATIONS:
Overall Officials: Candace L Ward, MD, MPH, Principal Investigator — Albert Einstein Medical Center Phialdelphia
Locations (2):
- United States (2):
  - Albert Einstein Medical Center Montgomery, East Norriton, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD with other researchers.

REFERENCES:
- [Background] 3M Critical and Chronic Care Solutions Division. 3M Steri-Strip Adhesive Skin Closures Application and Removal Pocket Guide. 3M Steri-Strip Adhesive Skin Closures Application and Removal Pocket Guide, 3M, 2013.
- [Background] Katz KH, Desciak EB, Maloney ME. The optimal application of surgical adhesive tape strips. Dermatol Surg. 1999 Sep;25(9):686-8. doi: 10.1046/j.1524-4725.1999.99084.x. PMID 10491057
- [Background] Rodeheaver GT, McLane M, West L, Edlich RF. Evaluation of surgical tapes for wound closure. J Surg Res. 1985 Sep;39(3):251-7. doi: 10.1016/0022-4804(85)90150-7. PMID 4033109
- [Background] Pushpakumar SB, Hanson RP, Carroll S. The application of Steri-Strips. Plast Reconstr Surg. 2004 Mar;113(3):1106-7. doi: 10.1097/01.prs.0000107747.92015.b7. No abstract available. PMID 15108939